CLINICAL TRIAL: NCT03056040
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study of ALXN1210 Versus Eculizumab in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Currently Treated With Eculizumab
Brief Title: ALXN1210 Versus Eculizumab in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH) Currently Treated With Eculizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-302; 2016-002026-36 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2019-03-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab; eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab (Experimental): On Day 1, participants received weight-based doses of ravulizumab ranging from 2400 to 3000 milligrams (mg). Thereafter, weight-based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Days 15, 71, and 127.
  After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants will receive weight-based doses of ravulizumab for up to 4 years.
  Interventions: Biological: Ravulizumab
- Eculizumab (Active Comparator): Participants received 900 mg of eculizumab every 2 weeks (q2w) for 26 weeks.
  After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants will receive weight-based doses of ravulizumab for up to 4 years.
  Interventions: Biological: Ravulizumab; Biological: Eculizumab

INTERVENTIONS:
Biological: Ravulizumab — All treatments were given as intravenous (IV) infusions. For participants weighing ≥40 to <60 kilograms (kg): 2400 mg was given as a single loading dose, followed by 3000 mg as maintenance dose. For participants weighing ≥60 to <100 kg: 2700 mg was given as a loading dose, followed by 3300 mg as maintenance dose. For participants weighing ≥100 kg: 3000 mg was given as a loading dose, followed by 3600 mg as maintenance dose.
  Other Names: ALXN1210; ULTOMIRIS
Biological: Eculizumab — All treatments were given as IV infusions. Participants received 900 mg of eculizumab q2w.
  Arms: Eculizumab

SUMMARY:
The primary purpose of this study was to assess the noninferiority of ravulizumab compared to eculizumab in adult participants with PNH who were clinically stable after having been treated with eculizumab for at least 6 months.

DETAILED DESCRIPTION:
The study consisted of a 4-week Screening Period and a 26-week Randomized Treatment Period (Primary Evaluation Period). After completion of the Primary Evaluation Period, all participants had the opportunity to enter the Extension Period, wherein participants will receive ravulizumab for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Treated with eculizumab for PNH for at least 6 months prior to Day 1.
3. Lactate dehydrogenase level ≤1.5 times the upper limit of normal (ULN) at screening.
4. PNH diagnosis confirmed by documented by high-sensitivity flow cytometry.
5. Documented meningococcal vaccination not more than 3 years prior to, or at the time of, initiating study treatment.
6. Female participants of childbearing potential must use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.
7. Willing and able to give written informed consent and comply with study visit schedule.

Exclusion Criteria:

1. History of bone marrow transplantation.
2. Body weight <40 kilograms at screening.
3. History of or ongoing major cardiac, pulmonary, renal, endocrine, or hepatic disease that, in the opinion of the investigator or sponsor, would preclude participation.
4. Unstable medical conditions (for example, myocardial ischemia, active gastrointestinal bleeding, severe congestive heart failure, anticipated need for major surgery within 6 months of randomization, or coexisting chronic anemia unrelated to PNH).
5. Female participants who are pregnant, breastfeeding, or who have a positive pregnancy test at screening or Day 1.
6. Participation in another interventional clinical study or use of any experimental therapy within 30 days before initiation of study treatment on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (5):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, The Bronx, New York
- Australia (5):
  - Research Site, Canberra
  - Research Site, Kogarah
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Woolloongabba
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (8):
  - Research Site, Amiens
  - Research Site, La Tronche
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
- Germany (3):
  - Research Site, Aachen
  - Research Site, Essen
  - Research Site, Ulm
- Italy (5):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Torino
  - Research Site, Vicenza
- Japan (5):
  - Research Site, Fukushima
  - Research Site, Kanazawa
  - Research Site, Shinagawa-ku
  - Research Site, Suita-shi
  - Research Site, Suwa-shi
- Netherlands (2):
  - Research Site, Maastricht
  - Research Site, Nijmegen
- South Korea (6):
  - Research Site, Bucheon-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
- United Kingdom (3):
  - Research Site, Airdrie
  - Research Site, Leeds
  - Research Site, London

REFERENCES:
- [Background] Kulasekararaj AG, Hill A, Rottinghaus ST, Langemeijer S, Wells R, Gonzalez-Fernandez FA, Gaya A, Lee JW, Gutierrez EO, Piatek CI, Szer J, Risitano A, Nakao S, Bachman E, Shafner L, Damokosh AI, Ortiz S, Roth A, Peffault de Latour R. Ravulizumab (ALXN1210) vs eculizumab in C5-inhibitor-experienced adult patients with PNH: the 302 study. Blood. 2019 Feb 7;133(6):540-549. doi: 10.1182/blood-2018-09-876805. Epub 2018 Dec 3. PMID 30510079
- [Background] Brodsky RA, Peffault de Latour R, Rottinghaus ST, Roth A, Risitano AM, Weitz IC, Hillmen P, Maciejewski JP, Szer J, Lee JW, Kulasekararaj AG, Volles L, Damokosh AI, Ortiz S, Shafner L, Liu P, Hill A, Schrezenmeier H. Characterization of breakthrough hemolysis events observed in the phase 3 randomized studies of ravulizumab versus eculizumab in adults with paroxysmal nocturnal hemoglobinuria. Haematologica. 2021 Jan 1;106(1):230-237. doi: 10.3324/haematol.2019.236877. PMID 31949012
- [Background] Ishiyama K, Nakao S, Usuki K, Yonemura Y, Ikezoe T, Uchiyama M, Mori Y, Fukuda T, Okada M, Fujiwara SI, Noji H, Rottinghaus S, Aguzzi R, Yokosawa J, Nishimura JI, Kanakura Y, Okamoto S. Results from multinational phase 3 studies of ravulizumab (ALXN1210) versus eculizumab in adults with paroxysmal nocturnal hemoglobinuria: subgroup analysis of Japanese patients. Int J Hematol. 2020 Oct;112(4):466-476. doi: 10.1007/s12185-020-02934-6. Epub 2020 Aug 31. PMID 32869125
- [Background] Kulasekararaj AG, Griffin M, Langemeijer S, Usuki K, Kulagin A, Ogawa M, Yu J, Mujeebuddin A, Nishimura JI, Lee JW, Peffault de Latour R; 301/302 Study Group. Long-term safety and efficacy of ravulizumab in patients with paroxysmal nocturnal hemoglobinuria: 2-year results from two pivotal phase 3 studies. Eur J Haematol. 2022 Sep;109(3):205-214. doi: 10.1111/ejh.13783. Epub 2022 Jun 16. PMID 35502600
- [Background] Kulasekararaj AG, Hill A, Langemeijer S, Wells R, Gonzalez Fernandez FA, Gaya A, Ojeda Gutierrez E, Piatek CI, Mitchell L, Usuki K, Bosi A, Brodsky RA, Ogawa M, Yu J, Ortiz S, Roth A, Lee JW, Peffault de Latour R. One-year outcomes from a phase 3 randomized trial of ravulizumab in adults with paroxysmal nocturnal hemoglobinuria who received prior eculizumab. Eur J Haematol. 2021 Mar;106(3):389-397. doi: 10.1111/ejh.13564. Epub 2021 Jan 3. PMID 33301613
- [Background] Peffault de Latour R, Brodsky RA, Ortiz S, Risitano AM, Jang JH, Hillmen P, Kulagin AD, Kulasekararaj AG, Rottinghaus ST, Aguzzi R, Gao X, Wells RA, Szer J. Pharmacokinetic and pharmacodynamic effects of ravulizumab and eculizumab on complement component 5 in adults with paroxysmal nocturnal haemoglobinuria: results of two phase 3 randomised, multicentre studies. Br J Haematol. 2020 Nov;191(3):476-485. doi: 10.1111/bjh.16711. Epub 2020 May 24. PMID 32449174
- [Background] Schrezenmeier H, Kulasekararaj A, Mitchell L, Sicre de Fontbrune F, Devos T, Okamoto S, Wells R, Rottinghaus ST, Liu P, Ortiz S, Lee JW, Socie G. One-year efficacy and safety of ravulizumab in adults with paroxysmal nocturnal hemoglobinuria naive to complement inhibitor therapy: open-label extension of a randomized study. Ther Adv Hematol. 2020 Oct 24;11:2040620720966137. doi: 10.1177/2040620720966137. eCollection 2020. PMID 33178408
- [Background] Wietz IC, Kulagin A, Nakao S, Piatek CI, Szer J, Rottinghaus ST, Volles L, Damokosh AI, Aguzzi R, Larratt L, Risitano AM. A Phase 3 study of ravulizumab (ALXN1210) versus eculizumab in adults with paroxysmal nocturnal hemoglobinuria naive to complement inhibitors: results of a subgroup analysis with patients stratified by baseline hemolysis level, transfusion history, and demographics. Blood. 2018;132 (Supplement 1):627. doi: 10.1182/blood-2018-99-110623
- [Derived] Kulasekararaj A, Brodsky R, Schrezenmeier H, Griffin M, Roth A, Piatek C, Ogawa M, Yu J, Patel AS, Patel Y, Notaro R, Usuki K, Kulagin A, Gualandro S, Fureder W, Peffault de Latour R, Szer J, Lee JW. Ravulizumab demonstrates long-term efficacy, safety and favorable patient survival in patients with paroxysmal nocturnal hemoglobinuria. Ann Hematol. 2025 Jan;104(1):81-94. doi: 10.1007/s00277-025-06193-5. Epub 2025 Jan 22. PMID 39841198
- [Derived] Schwartz CE, Stark RB, Borowiec K, Nolte S, Myren KJ. Norm-based comparison of the quality-of-life impact of ravulizumab and eculizumab in paroxysmal nocturnal hemoglobinuria. Orphanet J Rare Dis. 2021 Sep 15;16(1):389. doi: 10.1186/s13023-021-02016-8. PMID 34526067
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-PNH-302&attachmentIdentifier=c826be5c-044d-4dab-9e62-2d48684248c7&fileName=ALXN1210-PNH-302-CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified into 1 of 2 groups based on their transfusion history. Stratified participants were randomly assigned in a 1:1 ratio to receive ravulizumab or eculizumab.
Groups:
- Ravulizumab/Ravulizumab: On Day 1, participants received weight-based doses of ravulizumab ranging from 2400 to 3000 mg. Thereafter, weight- based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Days 15, 71, and 127. After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 4 years.
- Eculizumab/Ravulizumab: Participants received 900 mg of eculizumab every 2 weeks (q2w) for 26 weeks. After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 4 years.
Period: Primary Evaluation Period
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Started | 98 | 99
Received at Least 1 Dose of Study Drug (Participants included in the Safety Set) | 97 | 98
Participants in the Full Analysis Set (FAS) | 97 | 98
Completed | 96 | 95
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Randomized, not treated | 1 | 1
Period: Extension Period
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Started | 96 | 95
Completed | 92 | 88
Not Completed | 4 | 7
Not completed — Physician Decision | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study treatment (ravulizumab or eculizumab).
Groups:
- Eculizumab/Ravulizumab: Participants received 900 mg of eculizumab q2w for 26 weeks. After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 4 years.
- Total: Total of all reporting groups
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first infusion of study drug
  years | 46.6 (14.41) | 48.8 (13.97) | 47.7 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 97
  Male | 50 | 48 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 76 | 77 | 153
  Unknown or Not Reported | 18 | 17 | 35
Race/Ethnicity, Customized [Number; unit: participants]
  White | 50 | 61 | 111
  Asian | 23 | 19 | 42
  Not Reported | 13 | 13 | 26
  Black or African American | 5 | 3 | 8
  Unknown | 3 | 1 | 4
  Other | 2 | 1 | 3
  Multiple | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change In Lactate Dehydrogenase Levels From Baseline To Day 183
Description: Lactate dehydrogenase (LDH) is an indicator of intravascular hemolysis that occurs in participants with paroxysmal nocturnal hemoglobinuria. A decrease in LDH indicates reduction (improvement) in hemolysis. Baseline was defined as the average of all available on-study assessments prior to the first study drug infusion. The percent change in LDH was analyzed using a mixed-effect model for repeated measures (MMRM) with the fixed, categorical effects of treatment, study visit, and study visit by treatment group interaction, as well as the continuous, fixed covariate of baseline LDH and the stratification randomization indicator of packed red blood cells transfusion history (yes/no within 12 months prior to Day 1).
Time Frame: Baseline, Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Eculizumab/Ravulizumab: Participants who were randomized to the eculizumab group in the Primary Evaluation Period received a weight-based loading dose of ravulizumab on Day 183 followed by weight-based maintenance doses of ravulizumab 2 weeks later and q8w until the end of study (up to 4 years).
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 97 | 98
percent change | -0.82 [-7.75 to 6.11] | 8.39 [1.47 to 15.32]
Statistical Analysis 1: Comparison: Ravulizumab/Ravulizumab vs Eculizumab/Ravulizumab; Adjusting for a possible 10% dropout rate, a minimum of 192 participants were estimated to provide 90% power to demonstrate noninferiority of ravulizumab to eculizumab; Test type: Non-Inferiority — A difference in percent change in LDH between the ravulizumab and eculizumab treatment groups at Day 183 along with a 2-sided 95% confidence interval (CI) was calculated. Noninferiority margin (NIM) was based on the upper bound of the 95% CI. NIM was 15%; Treatment Difference = -9.21, 95% CI 2-sided [-18.84 to 0.42] — Treatment difference was estimated for ravulizumab - eculizumab

2. Secondary Outcome: Number Of Participants With Breakthrough Hemolysis Through Day 183
Description: Breakthrough hemolysis (BTH) was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, dyspnea, anemia [hemoglobin <10 grams (g)/deciliter (dL)], major adverse vascular event [including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2 times the upper limit of normal (ULN).
Time Frame: Baseline through Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab).
Measure: Number (95% Confidence Interval); unit: number of participants
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 97 | 98
number of participants | 0 [0.00 to 3.73] | 5 [1.68 to 11.51]
Statistical Analysis 1: Comparison: Ravulizumab/Ravulizumab vs Eculizumab/Ravulizumab; A difference in the percentages of participants with BTH was calculated between the ravulizumab and eculizumab treatment groups, along with a 95% CI for the difference using the stratified Newcombe CI method. The stratification factor observed was transfusion history within 1 year prior to first dose of study drug; Test type: Non-Inferiority — NIM was based on the upper bound of the 95% CI. NIM was 20%; Treatment Difference = -5.1, 95% CI 2-sided [-18.99 to 8.89] — Treatment difference was estimated for ravulizumab - eculizumab

3. Secondary Outcome: Change From Baseline To Day 183 In Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Scores
Description: FACIT-Fatigue score ranges from 0 to 52, with a higher score indicating less fatigue. Baseline was defined as the last non-missing assessment value prior to first study drug dose. Change in FACIT-Fatigue score from Baseline to Day 183 was analyzed using an MMRM with the fixed, categorical effects of treatment, the stratification randomization indicator of packed red blood cells transfusion history (yes/no within 12 months prior to Day 1), study visit, and study visit by treatment group interaction, as well as the continuous fixed covariate of Baseline FACIT-Fatigue score.
Time Frame: Baseline, Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 97 | 98
units on a scale | 2.01 [0.64 to 3.39] | 0.54 [-0.84 to 1.93]
Statistical Analysis 1: Comparison: Ravulizumab/Ravulizumab vs Eculizumab/Ravulizumab; Test type: Non-Inferiority — NIM was based on the lower bound of the 95% CI. NIM margin was -3; Treatment Difference = 1.47, 95% CI 2-sided [-0.21 to 3.15] — Treatment difference was estimated for ravulizumab - eculizumab

4. Secondary Outcome: Percentage Of Participants Who Achieved Transfusion Avoidance Through Day 183
Description: Transfusion avoidance was defined as the percentage of participants who remained transfusion free and did not require a transfusion per protocol-specified guidelines (hemoglobin value of ≤9 g/dL with signs or symptoms of sufficient severity to warrant a transfusion, or a hemoglobin value of ≤7 g/dL regardless of presence of clinical signs or symptoms) through Day 183.
Time Frame: Baseline through Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 97 | 98
percentage of participants | 87.6 [81.08 to 94.18] | 82.7 [75.16 to 90.15]
Statistical Analysis 1: Comparison: Ravulizumab/Ravulizumab vs Eculizumab/Ravulizumab; A difference in the percentages of participants achieving transfusion avoidance was calculated between the ravulizumab and eculizumab treatment groups, along with a 95% CI for the difference using the stratified Newcombe CI method. The stratification factor observed was transfusion history within 1 year prior to first dose of study drug; Test type: Non-Inferiority — NIM was based on the lower bound of the 95% CI. NIM was -20%; Treatment Difference = 5.5, 95% CI 2-sided [-4.27 to 15.68] — Treatment difference was estimated for ravulizumab - eculizumab

5. Secondary Outcome: Percentage Of Participants With Stabilized Hemoglobin Levels Through Day 183
Description: Stabilized hemoglobin was defined as avoidance of a ≥2 g/dL decrease in hemoglobin level from Baseline in the absence of transfusion through Day 183.
Time Frame: Baseline through Day 183
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 97 | 98
percentage of participants | 76.3 [67.82 to 84.75] | 75.5 [67.00 to 84.02]
Statistical Analysis 1: Comparison: Ravulizumab/Ravulizumab vs Eculizumab/Ravulizumab; A difference in the percentages of participants with stabilized hemoglobin was calculated between the ravulizumab and eculizumab treatment groups, along with a 95% CI for the difference using the stratified Newcombe CI method. The stratification factor observed was transfusion history within 1 year prior to first dose of study drug; Test type: Non-Inferiority — NIM was based on the lower bound of the 95% CI. NIM was -20%; Treatment Difference = 1.4, 95% CI 2-sided [-10.41 to 13.31] — Treatment difference was estimated for ravulizumab - eculizumab

6. Secondary Outcome: Number Of Participants With Breakthrough Hemolysis Through End of Study
Description: BTH was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, dyspnea, anemia [hemoglobin <10 g/dL], major adverse vascular event [including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2 times the ULN.
Time Frame: Baseline through end of study (up to 4 years)
Population: Full Analysis Set: All participants who received at least 1 dose of randomized treatment (ravulizumab or eculizumab). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: number of participants
Groups:
- Ravulizumab/Ravulizumab: Participants who were randomized to the ravulizumab group in the Primary Evaluation Period continued to receive maintenance doses of ravulizumab every 8 weeks (q8w) until the end of study (up to 4 years).
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 96 | 95
number of participants | 9 [4.38 to 17.05] | 6 [2.35 to 13.24]

7. Secondary Outcome: Change From Baseline To End of Study In FACIT-Fatigue Scores Through End of Study
Description: as for outcome 3
Time Frame: Baseline, End of Study (up to 4 years)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ravulizumab/Ravulizumab: Participants who were randomized to the ravulizumab group in the Primary Evaluation Period continued to receive maintenance doses of ravulizumab q8w until the end of study (up to 4 years)
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 14 | 13
units on a scale | -1.43 (5.694) | 0.00 (5.944)

8. Secondary Outcome: Percentage Of Participants Who Achieved Transfusion Avoidance Through End of Study
Description: Transfusion avoidance was defined as the percentage of participants who remained transfusion free and did not require a transfusion per protocol-specified guidelines (hemoglobin value of ≤9 g/dL with signs or symptoms of sufficient severity to warrant a transfusion, or a hemoglobin value of ≤7 g/dL regardless of presence of clinical signs or symptoms) through the end of study.
Time Frame: Baseline through end of study (up to 4 years)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 96 | 95
percentage of participants | 70.83 [60.67 to 79.67] | 70.53 [60.29 to 79.44]

9. Secondary Outcome: Percentage Of Participants With Stabilized Hemoglobin Levels Through End of Study
Description: Stabilized hemoglobin was defined as avoidance of a ≥2 g/dL decrease in hemoglobin level from Baseline in the absence of transfusion through end of study.
Time Frame: Baseline through end of study (up to 4 years)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab/Ravulizumab | Eculizumab/Ravulizumab
Number analyzed (Participants) | 96 | 95
percentage of participants | 58.33 [47.82 to 68.32] | 67.37 [59.68 to 76.64]

ADVERSE EVENTS:
Time Frame: From Baseline (after first dose) to end of study (up to 4 years)
Description: Primary Evaluation Period (26 weeks)- Ravulizumab Treatment: data for All-Cause Mortality, Serious Adverse Events, and Other Adverse Events are for participants in the Ravulizumab-Treated Set. Eculizumab Treatment: data for All-Cause Mortality, Serious Adverse Events, and Other Adverse Events are for the participants in the Safety Set. Extension Period-data for All-Cause Mortality, Serious Adverse Events, and Other Adverse Events are for the participants in the Ravulizumab-Treated Set.
Groups:
- Primary Evaluation Period (26 Weeks) Ravulizumab Treatment: On Day 1, participants received weight- based doses of ravulizumab ranging from 2400 to 3000 mg. Thereafter, weight- based doses of ravulizumab ranging from 3000 to 3600 mg were administered on Days 15, 71, and 127.
- Primary Evaluation Period (26 Weeks) Eculizumab Treatment: Participants received 900 mg of eculizumab q2w for 26 weeks.
- Extension Period (Ravulizumab To Ravulizumab); Extension Period (Eculizumab to Ravulizumab): After completion of the 26-week Primary Evaluation Period, participants had the opportunity to enter the Extension Period, wherein participants received weight-based doses of ravulizumab for up to 4 years.
Arm/Group | Primary Evaluation Period (26 Weeks) Ravulizumab Treatment | Primary Evaluation Period (26 Weeks) Eculizumab Treatment | Extension Period (Ravulizumab To Ravulizumab) | Extension Period (Eculizumab to Ravulizumab)
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/96 | 3/95
Serious Adverse Events (participants affected / at risk) | 4/97 | 8/98 | 26/96 | 33/95
Other Adverse Events (participants affected / at risk) | 72/97 | 85/98 | 83/96 | 85/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Evaluation Period (26 Weeks) Ravulizumab Treatment (N=97) | Primary Evaluation Period (26 Weeks) Eculizumab Treatment (N=98) | Extension Period (Ravulizumab To Ravulizumab) (N=96) | Extension Period (Eculizumab to Ravulizumab) (N=95)
Haemolysis (Blood and lymphatic system disorders) | 0 | 2 | 1 | 4
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 5 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cerebrospinal fluid retention (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Evaluation Period (26 Weeks) Ravulizumab Treatment (N=97) | Primary Evaluation Period (26 Weeks) Eculizumab Treatment (N=98) | Extension Period (Ravulizumab To Ravulizumab) (N=96) | Extension Period (Eculizumab to Ravulizumab) (N=95)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 7 | 9 | 12 | 11
Constipation (Gastrointestinal disorders) | 6 | 5 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 7 | 15 | 14
Nausea (Gastrointestinal disorders) | 8 | 9 | 13 | 16
Vomiting (Gastrointestinal disorders) | 6 | 4 | 7 | 4
Chest pain (General disorders) | 3 | 9 | 5 | 5
Fatigue (General disorders) | 7 | 6 | 18 | 19
Influenza like illness (General disorders) | 6 | 8 | 9 | 9
Pyrexia (General disorders) | 9 | 2 | 15 | 16
Nasopharyngitis (Infections and infestations) | 20 | 20 | 27 | 21
Rhinitis (Infections and infestations) | 5 | 4 | 10 | 7
Upper respiratory tract infection (Infections and infestations) | 19 | 10 | 24 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 11
Dizziness (Nervous system disorders) | 3 | 7 | 8 | 15
Headache (Nervous system disorders) | 27 | 17 | 21 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 16 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 8 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 7 | 10
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 7 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 6 | 5
Urinary tract infection (Infections and infestations) | 1 | 0 | 7 | 8
Gastroenteritis (Infections and infestations) | 1 | 0 | 7 | 3
Influenza (Infections and infestations) | 1 | 0 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 10 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 11 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 5
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 5 | 4
Oedema peripheral (General disorders) | 0 | 0 | 5 | 4
Asthenia (General disorders) | 0 | 0 | 5 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 5
COVID-19 (Infections and infestations) | 0 | 0 | 5 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 5
Infection (Infections and infestations) | 0 | 0 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 2
Migraine (Nervous system disorders) | 0 | 0 | 3 | 5
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Viral infection (Infections and infestations) | 0 | 0 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03056040/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03056040/SAP_001.pdf